CLINICAL TRIAL: NCT05233267
Title: Neopterin on Admission to the ICU: an Immunological Biomarker That Could Help Admission Decisions by Identifying Elderly Patients (≥80 Years) Able to Survive an ICU Stay Without Disability
Brief Title: Neopterin on Admission to Intensive Care Unit
Acronym: NUAGE
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: APHP210083; 2021-A02264-37 (Registry Identifier: DRCB)
Record Dates: First submitted 2022-02-09; First posted 2022-02-10 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Elderly Patient (80 Years Old or More) Admitted to Intensive Care
Keywords: neopterin
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Blood sample — Dosage of neopterin

SUMMARY:
For the last twenty years, the proportion of patients aged 80 years and more, hospitalized in intensive care (ICU) has been increasing. The question of the admission of an elderly patient in intensive care raises many medico-socio-economic questions. The general objective of geriatric management is to improve the survival of the patient by maintaining his autonomy. Before an invasive management, it is therefore important to assess which patients are capable of surviving in good conditions. Moreover, as intensive care resources are not extensible, it is important to rationalise the use of this type of care. To date, there are no reliable criteria for predicting which patients will benefit from ICU care. The use of a predictive biomarker, in addition to the existing scores which are not very effective in this population, could guide the intensive care physician in his decision which is generally made in the emergency.

The hypothesis of the study is that neopterin measured on admission of the elderly patient to the ICU may improve prediction of survival without major loss of autonomy at 3 months. Acute stress induced by a serious pathology has a profound impact on the immune system via the activation of the neuroendocrine system and the production of endogenous cortisol. Usually, cortisol inhibits the production of pro-inflammatory cytokines such as interferon gamma (IFNg). Sometimes this inhibition is ineffective and leads to an intense pro-inflammatory state that is harmful to the body. Neopterin is produced by monocytes/macrophages under the influence of IFNg. It is associated with a poor prognosis in many diseases such as sepsis or cancer. In the comorbid elderly patient with an upper femoral fracture, the pre-operative neopterin level is predictive of one-year mortality and functional recovery.

The hypothesis of the study is that neopterin measured on admission of the elderly patient to the ICU may improve prediction of survival without major loss of autonomy at 3 months.

Each patient will be included on admission to the intensive care unit within a maximum of 24 hours (D0). Demographic data (age, sex), severity (IGSIII), comorbidity (CIRS), autonomy (ADL and IADL) and frailty (CFS) scores will be collected as well as the diagnosis at admission.

Two additional tubes will be collected during the entry assessment (performed as part of usual care) at inclusion (D0) for neopterin and other biomarkers (4 ml dry tube and 10 ml lithium heparin tube). The blood tubes will be transferred to the research laboratory within 48 hours after sampling. The determination of neopterin, cytokines and oxidative stress biomarkers will be performed by an enzyme-linked immunosorbent assay (Neopterin ELISA Kit CE-IVD, Tecan laboratory) at the Centre d'Immunologie et des Maladies Infectieuses (CIMI-Paris).

The assays will be performed at the end of the study, blinded to the patient's outcome, and the follow-up of the patients will be performed blinded to the results of the neopterin assay and the other markers.

Patients will be followed up at 3 months from inclusion (M3). The follow-up data will be collected during a routine geriatric consultation. During this consultation, the scores of comorbidities (CIRS), autonomy (ADL and IADL) and frailty (CFS) will be collected. An assessment of physical performance will be carried out by measuring the Short Physical Performance Battery (SPPBS) and the "Handgrip". If it is impossible to carry out the consultation (patient unable to move), the follow-up data (CIRS, ADL and CFS) will be collected from the patient or his relatives during a phone interview conducted by a clinical research technician.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 80 years old
* Admission to intensive care unit before 24 hours
* Non opposition expressed by the participant or its relative/trusty person, or emergency inclusion procedure

Exclusion Criteria:

* Hospitalisation for a scheduled surgery
* New admission within a month before previous stay to intensive care unit
* Active solid cancer or malignant hemopathy
* Immunosuppressant treatment (including corticotherapy > 5 mg/d)
* Autoimmune disease
* Tutorship or curatorship

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The population is selected from 80-year-old patients or more attending intensive care unit for less than 24 hours.
Sampling Method: Non-Probability Sample
Enrollment: 326 (Estimated)
Dates: Start 2022-11-21 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Survival without significant loss of autonomy | Month 3
  Autonomy is evaluated by Activities of Daily Living score (ADL). This score is based on a 6-item questionnaire. Each item is rated 0, 0.5 or 1. 1 is the best outcome.
  A significant loss of autonomy is defined by a ADL score at 3 month after inclusion lower by more than 1 point compared to the ADL score before hospitalization.

SECONDARY OUTCOMES:
Intra-hospital mortality | Month 3
Mortality | Month 3
Functional autonomy | Month 3
  Instrumental Activities of Daily Living score (IADL).This score is based on a 4-item questionnaire. Each item is rated 0 or 1. 1 is the best outcome.
Short Physical Performance Battery | Month 3
  The score is from 0 to 12 based on the result of three exercises: Balance, gait speed and chair stand. 12 means better outcome.
Handgrip test | Month 3
Neopterin | Day 0
  The concentration of neopterin is measured in blood.

OTHER OUTCOMES:
Simplified Acute Physiology Score III (SAPS3) | Day 0
  The score is based on 29-item questionnaire. The questionnaire is rated from 1 to 189, with 189 being the worst score. The final score is converted into a prognostic mortality score in percent.
Clinical Frailty Scale (CFS) | Day 0
  The scale is rated from 1 to 9, with 9 being the worst score.
Cumulative Illness Rating Scale (CIRS) | Day 0
  The scale is based on a 14-item questionnaire. Each item is rated from 0 to 4, with 4 being the worst score. The total score corresponds to the sum of the 14 items score.

CONTACTS AND LOCATIONS:
Overall Officials: Hélène VALLET, MD, Principal Investigator — Hôpital Saint-Antoine - APHP
Locations (1):
- Hôpital Saint-Antoine / Service de réanimation, Paris, France